CLINICAL TRIAL: NCT01461486
Title: Effectiveness of Continuous Positive Airway Pressure and Oral Appliances in Mild Obstructive Sleep Apnea: a Randomized, Parallel, Single Blind and Controlled Study
Brief Title: Continuous Positive Airway Pressure and Oral Appliances Treatments in Mild Obstructive Sleep Apnea
Acronym: OSAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Principal Investigator, Prof. Dr. Lia Azeredo-Bittencourt, Professor, Associação Fundo de Incentivo à Pesquisa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1300/11
Record Dates: First submitted 2011-10-25; First posted 2011-10-28 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Mild Obstructive Sleep Apnea Syndrome
Keywords: Continuous positive airway pressure; Oral appliance; mild Obstructive Sleep Apnea Syndrome
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Continuous Positive Airway Pressure (Active Comparator): Intervention group
  Interventions: Device: Continuous Positive Airway Pressure (CPAP)
- Oral Appliance (BRD) (Active Comparator): Intervention group
  Interventions: Device: Oral Appliance (BRD)
- Hygiene sleep care (No Intervention): Control group

INTERVENTIONS:
Device: Continuous Positive Airway Pressure (CPAP) — The device is a flow generator used to open the airway during sleep.
  Other Names: Resmed (trademark). Autoset Vantage - fixed pressure.
  Arms: Continuous Positive Airway Pressure
Device: Oral Appliance (BRD) — The device increases the volume of the airway by mandibular traction.
  Other Names: Brazilian Dental Appliance (BRD).
  Arms: Oral Appliance (BRD)

SUMMARY:
Treatment response of mild obstructive sleep apnea (OSA) to continuous positive airway pressure (CPAP) therapy and oral appliance (OA) is still controversial. The aim of this study is to evaluate the effect of CPAP and OA treatment on: objective and subjective sleepiness, cognitive deficits, mood changes, quality of life, inflammatory profile and metabolic cardiovascular and hormonal alterations in mild OSA subjects. Subjects with mild OSA (apnea -hypopnea index of 5 or more events per hour of sleep and less than 15), both genders, body mass index lower than 35Kg/m2 and age between 18 to 65 years will be included. They also must have a minimum mandibular protrusion of 7mm. Subjects will be randomly distributed in three groups: group 1 with CPAP, group 2 with OA and group 3 will be the control. At baseline evaluation, six months, one year and three years, all subjects will be submitted to sleep questionnaires, physical examination, ear-nose and throat evaluation, baseline polysomnography (and with CPAP for groups 1), Epworth Sleepiness Scale, Karolinska Sleepiness Scale, Stanford Sleepiness Scale, Maintenance of Wakefulness Test, Chalder Fatigue Scale, Neurocognitive testing, Beck Inventories of anxiety and depression, Functional Outcomes of Sleep Questionnaire (FOSQ), WHOQOL-BREF quality of life questionnaire, Short Form-36 quality of life questionnaire, questionnaire for sexual dysfunction, blood analysis for inflammatory, metabolic and hormonal evaluation, assessment of heart rate variability, 24 hour blood pressure monitoring and endothelial dysfunction. Sleep hygiene care was offer to three groups. Analysis mean and standard deviation will be used for descriptive statistical and a general linear model will be applied for analysis within groups on different time.

ELIGIBILITY:
Inclusion Criteria:

* Both genders;
* body mass index lower than 35Kg/m2;
* age between 18 and 65 years old;
* polysomnographic and clinical diagnosis of mild apnea (apnea-hypopnea index of 5 or more events per hour of sleep and less than 15 and minimum mandibular protrusion of 7mm.

Exclusion Criteria:

* Unsatisfactory dental conditions (active periodontal disease, extensive caries or insufficient teeth for appliance content);
* temporomandibular disorders (chronic joint or muscle disease); central apnea; claustrophobia and severe otorhinolaryngologic diseases (severe nasal septal deviation, marked hypertrophy of nasal turbinates, hypertrophy of tonsils and/or adenoids sharp);
* excessive use of alcohol and psychoactive drugs;
* clinical, neurological or psychiatric decompensated diseases;
* others sleep diseases and previous obstructive sleep apnea treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2011-10; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Excessive Daytime Sleepiness | From the baseline evaluation to three years after the treatment with continuous positive airway pressure and appliance oral.

SECONDARY OUTCOMES:
Evaluations of fatigue. | From the baseline evaluation to three years after the treatment with continuous positive airway pressure and appliance oral
Evaluation of cognition. | From the baseline evaluation to three years after the treatment with continuous positive airway pressure and appliance oral.
  Performance Vigilance Test (PVT)
Evaluation of depression. | From the baseline evaluation to three years after the treatment with continuous positive airway pressure and appliance oral.
  Beck Depression Inventory - BDI
Evaluation of quality of life. | From the baseline evaluation to three years after the treatment with continuous positive airway pressure and appliance oral
Evaluation of inflammation. | From the baseline evaluation to three years after the treatment with continuous positive airway pressure and appliance oral
  Blood analysis for inflammatory.
Evaluation of blood pressure. | From the baseline evaluation to three years after the treatment with continuous positive airway pressure and appliance oral
  Assessment of heart rate variability, 24 hour blood pressure monitoring and endothelial dysfunction.
Evaluation of sexual dysfunction. | From the baseline evaluation to three years after the treatment with continuous positive airway pressure and appliance oral
Evaluation of anxiety | From the baseline evaluation to three years after the treatment with continuous positive airway pressure and appliance oral
  Beck Anxiety Inventory - BAI
Evaluation of metabolism | From the baseline evaluation to three years after the treatment with continuous positive airway pressure and appliance oral
  Blood analysis for metabolism
Evaluation of hormonal alterations. | From the baseline evaluation to three years after the treatment with continuous positive airway pressure and appliance oral.
  Blood analysis for hormonal alterations.
Evaluation of heart rate variability | From the baseline evaluation to three years after the treatment with continuous positive airway pressure and appliance oral.
  Assessment of heart rate variability.
Evaluation of endothelial disfunction. | From the baseline evaluation to three years after the treatment with continuous positive airway pressure and appliance oral.
  Assessment of endothelial disfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Associação Fundo de Incentivo à Pesquisa, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Guimaraes TM, Poyares D, Oliveira E Silva L, Luz G, Coelho G, Dal Fabbro C, Tufik S, Bittencourt L. The treatment of mild OSA with CPAP or mandibular advancement device and the effect on blood pressure and endothelial function after one year of treatment. J Clin Sleep Med. 2021 Feb 1;17(2):149-158. doi: 10.5664/jcsm.8822. PMID 32964829
- [Derived] M Guimaraes T, Bittencourt L, P Luz G, O Silva L, Burke P, Coelho G, Milani A, Badke L, Togeiro S, Tufik S, Poyares D. Association between nondipping pattern and EndoPAT signal in patients with mild obstructive sleep apnea. Sleep Med. 2018 Nov;51:9-14. doi: 10.1016/j.sleep.2018.05.041. Epub 2018 Jun 27. PMID 30077018